CLINICAL TRIAL: NCT00665067
Title: Correlative Biomarker Study for MPD-RC Treatment Studies in the Philadelphia Chromosome Negative MPD
Brief Title: Correlative Biomarker Study in Patients With Myeloproliferative Disorders
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 07-0548-00107; P01CA108671-05 (NIH); MPD-RC 107 (Other: Myeloproliferative Disorders-Research Consortium)
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Myeloproliferative Disease; Myelofibrosis; Idiopathic Myelofibrosis; Essential Thrombocythemia; Polycythemia Vera
Keywords: Myeloproliferative Disease; Myelofibrosis; Idiopathic Myelofibrosis; Essential Thrombocythemia; Polycythemia Vera; Biomarkers; Philadelphia Chromosome Negative; Clonal Hematopoietic malignancies
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Leftover tissue will be asked for to be stored in the MPD-RC Tissue Bank
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Researchers will use abnormal blood and/or bone marrow cells, or materials derived from these abnormal cells, like DNA, RNA, protein or plasma, in laboratory studies. Toenail clippings will provide normal material like DNA for comparison with the abnormal material derived from the blood and/or bone marrow. The results of these studies will be correlated with subjects' disease symptoms and response to their experimental treatment. The MPD-RC researchers are interested in studying molecules from the blood and bone marrow, the exact molecules changing over time with the investigators choosing only the most promising for investigation.

The investigators are attempting to better understand the causes of MPD and to develop improved methods for the diagnosis and treatment of these diseases. These syndromes carry a high risk of developing leukemia. It is important to continue to learn more about these blood cancers and to learn more about the effectiveness and potential side effects of various treatments. It is believed that further basic knowledge about these cancer cells as well as the effects of treatment will lead to the improvement of current therapies and the development of entirely new treatments for these diseases. The MPD-RC is hoping to determine if a number of laboratory tests (biomarkers) will allow for the prediction of response in future patients to the treatment they would receive.

ELIGIBILITY:
Inclusion Criteria:

* Patients are to be registered to this study if they meet the eligibility criteria for one of the MPD-RC treatment protocols linked to this study.
* Patients diagnosed with the following Myeloproliferative disorders including: polycythemia vera (PV), idiopathic myelofibrosis (IM), and essential thrombocythemia (ET) who are participating in treatment protocols of the MPD-RC are eligible.
* Patients must have signed an informed consent to participate in a Myeloproliferative Disorders Research Consortium (MPD-RC) treatment study to which this protocol is a companion study. The subject must also have signed a consent to participate in this mandatory companion study.

Exclusion Criteria:

See inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in MPD-RC treatment protocols.
Sampling Method: Non-Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2007-04; Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
To collect and store tissue samples from patients with myeloproliferative disorders (PV,IM,and ET). Tissue samples will be used to perform a variety of biomarker studies to monitor the effects of a particular therapeutic intervention. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Rona S Weinberg, PhD, Study Chair — Myeloproliferative Disorders-Research Consortium; John Mascarenhas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (22):
- United States (15):
  - Mayo Clinic, Scottsdale, Arizona
  - The Palo Alto Clinic, Palo Alto, California
  - Georgetown University, Washington D.C., District of Columbia
  - Emory Hospital, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical College, New York, New York
  - New York Blood Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Geisinger Cancer Center, Hazleton, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Italy (5):
  - Ospedali Riuniti di Bergamo, Bergamo
  - University of Florence, Florence
  - Ospedale San Martino Genova, Genova
  - San Matteo Hospital, Pavia
  - Universita Cattolica del Sacro Cuore, Rome
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom